CLINICAL TRIAL: NCT06307860
Title: Comparison of Pulse Field Ablation and Radiofrequency Ablation in Left Atrial Reverse Remodeling in Patients With Paroxysmal Atrial Fibrillation
Brief Title: Comparison of Different Ablation Surgeries on Left Atrial Reverse Remodeling in Patients With Atrial Fibrillation
Status: Recruiting | Type: Observational
Sponsor: Yun Wan (Other)
Responsible Party: Sponsor-Investigator, Yun Wan, resident doctor, The Affiliated Ganzhou Hospital of Nanchang University
Organization: The Affiliated Ganzhou Hospital of Nanchang University (Other)
Other Study IDs: 15270977512@163.com
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation
Keywords: Pulsed field ablation; radiofrequency ablation; atrial fibrillation; reconfiguration
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- P group: Perform pulsed field ablation surgery after meeting the inclusion criteria
  Interventions: Device: pulsed field ablation
- R group: Perform radiofrequency ablation surgery after meeting the inclusion criteria
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Device: pulsed field ablation — Selected patients were selected to undergo relevant surgeries, and their preoperative and postoperative baseline data were collected. They were followed up for 6 months after surgery.
  Groups: P group
Procedure: radiofrequency ablation — Selected patients were selected to undergo relevant surgeries, and their preoperative and postoperative baseline data were collected. They were followed up for 6 months after surgery.
  Groups: R group

SUMMARY:
The goal of this Ambispective cohort Study is to compare in patients with paroxysmal atrial fibrillation undergo pulse field ablation and radiofrequency ablation, respectively. The main question it aims to answer are:Comparison of the therapeutic effects of pulse field ablation and traditional thermal ablation on patients with paroxysmal atrial fibrillation and postoperative left atrial reverse remodeling.Participants will Perform pulse field ablation or radiofrequency ablation according to different groups, and cooperate to complete outpatient follow-up 6 months after surgery.

DETAILED DESCRIPTION:
Patients with paroxysmal atrial fibrillation who underwent ablation surgery at Ganzhou People's Hospital from June 2022 to June 2024 were divided into two groups: pulse ablation group (P group) and radiofrequency ablation group (R group). Collect baseline data, preoperative and postoperative heart rate, white blood cell count, neutrophil to lymphocyte ratio, and uric acid, evaluate and record surgical data and postoperative complications for both groups, and follow up for 6 months after discharge. Collect and analyze the recurrence rate of atrial arrhythmias, electrocardiogram, echocardiography, and left atrial CTA of patients. Compare surgical data, postoperative complications, atrial structure and function, P-wave dispersion, and pulmonary vein stenosis between two groups.

ELIGIBILITY:
Inclusion Criteria:

* 1.Aged between 18-75 years old; 2.Patients confirmed by electrocardiogram or clinically diagnosed with atrial fibrillation; 3.Atrial fibrillation that terminates spontaneously or through intervention within 7 days after onset; 4.Accompanied by symptoms of atrial fibrillation; 5.The patient has a willingness to undergo catheter ablation treatment; 6.The patient agrees to be enrolled and has high compliance. They voluntarily participate in the trial, sign an informed consent form, and cooperate with the follow-up of this project.

Exclusion Criteria:

* 1.The echocardiography shows that the anterior posterior diameter of the left atrium is ≥ 50mm, and the LVEF is ≤ 40%; 2.Esophageal echocardiography or CT examination suggests thrombus in the left atrium/left atrial appendage; 3.Preoperative confirmation of typical atrial flutter or other supraventricular tachycardia by electrocardiogram or Holter; 4.Previously underwent catheter ablation or other surgeries due to atrial fibrillation; 5.Previously underwent left atrial appendage closure surgery or left atrial appendage closure surgery, or planned to undergo one-stop left atrial appendage closure surgery; 6.Previously underwent valve repair or valve replacement surgery; 7.Implantable metal cardiac instruments that have implanted pacemakers, implantable cardioverters, defibrillators, or other devices that may interfere with the energy field of pulsed electric field ablation; 8.New York Heart Function Classification (NYHA) Level III or IV; 9.Cardiovascular events within 3 months prior to surgery (including acute myocardial infarction, coronary intervention or bypass surgery, atrial or ventricular incision); 10.Has undergone any carotid stent implantation or endarterectomy within 6 months prior to surgery; 11.Thromboembolic events (including transient ischemic attacks) occurring within 6 months prior to surgery; 12.Existence of wall thrombus, atrial septal occluder or patch, tumor, myxoma, or other abnormal conditions that hinder vascular puncture or catheter operation; 13.Severe lung disease (such as restrictive lung disease, constrictive or chronic obstructive pulmonary disease) or any other lung or respiratory system disease or dysfunction that can cause severe chronic symptoms; 14.Atrial fibrillation secondary to electrolyte disorders, thyroid diseases, or other reversible causes; 15.Known pulmonary vein stenosis; 16;Systemic active infection; 17.Severe organic heart disease; 18.Contraindications to anticoagulant therapy, X-rays, and severe hematological disorders; 19.Expected life<12 months; 20.Pregnancy test positive for women of childbearing age or in lactation or planning to conceive within the next 12 months; 21.Patients who are participating in clinical trials of other experimental biological agents, drugs, or devices and have not completed them; 22.Other researchers believe that it is not appropriate to participate in this experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion of paroxysmal atrial fibrillation patients who underwent ablation surgery at Ganzhou People's Hospital between June 2022 and June 2024 and met the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of atrial arrhythmias | Follow up for 6 months after surgery
  Follow up patients for any recurrent symptoms and recheck electrocardiograms for atrial arrhythmias
Left atrial end diastolic diameter | Follow up for 6 months after surgery
  Follow up patient's left atrial diastolic diameter indicated by echocardiography and left atrial CTA

SECONDARY OUTCOMES:
p wave dispersion | Follow up for 6 months after surgery
  ECG measurement of P-wave dispersion
Pulmonary vein stenosis rate | Follow up for 6 months after surgery
  Pulmonary vein CTA assessment of pulmonary vein stenosis

OTHER OUTCOMES:
Postoperative complications | Complete surgery until 6 months after surgery
  Evaluate the occurrence of complications after completing ablation surgery

CONTACTS AND LOCATIONS:
Overall Officials: Wan Yun, Bachelor, Study Director — The Affiliated Ganzhou Hospital, Jiangxi Medical College, Nanchang University
Locations (1):
- Ganzhou People's Hospital, Ganzhou, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided
At present, complete data has not been obtained

REFERENCES:
- [Result] Lloyd-Jones DM, Wang TJ, Leip EP, Larson MG, Levy D, Vasan RS, D'Agostino RB, Massaro JM, Beiser A, Wolf PA, Benjamin EJ. Lifetime risk for development of atrial fibrillation: the Framingham Heart Study. Circulation. 2004 Aug 31;110(9):1042-6. doi: 10.1161/01.CIR.0000140263.20897.42. Epub 2004 Aug 16. PMID 15313941
- [Result] Du X, Guo L, Xia S, Du J, Anderson C, Arima H, Huffman M, Yuan Y, Zheng Y, Wu S, Guang X, Zhou X, Lin H, Cheng X, Dong J, Ma C. Atrial fibrillation prevalence, awareness and management in a nationwide survey of adults in China. Heart. 2021 Jan 28;107(7):535-41. doi: 10.1136/heartjnl-2020-317915. Online ahead of print. PMID 33509976
- [Result] Heijman J, Voigt N, Nattel S, Dobrev D. Cellular and molecular electrophysiology of atrial fibrillation initiation, maintenance, and progression. Circ Res. 2014 Apr 25;114(9):1483-99. doi: 10.1161/CIRCRESAHA.114.302226. PMID 24763466
- [Result] Igarashi T, Finet JE, Takeuchi A, Fujino Y, Strom M, Greener ID, Rosenbaum DS, Donahue JK. Connexin gene transfer preserves conduction velocity and prevents atrial fibrillation. Circulation. 2012 Jan 17;125(2):216-25. doi: 10.1161/CIRCULATIONAHA.111.053272. Epub 2011 Dec 8. PMID 22158756
- [Result] Camm AJ, Naccarelli GV, Mittal S, Crijns HJGM, Hohnloser SH, Ma CS, Natale A, Turakhia MP, Kirchhof P. The Increasing Role of Rhythm Control in Patients With Atrial Fibrillation: JACC State-of-the-Art Review. J Am Coll Cardiol. 2022 May 17;79(19):1932-1948. doi: 10.1016/j.jacc.2022.03.337. PMID 35550691
- [Result] Noubiap JJ, Feteh VF, Middeldorp ME, Fitzgerald JL, Thomas G, Kleinig T, Lau DH, Sanders P. A meta-analysis of clinical risk factors for stroke in anticoagulant-naive patients with atrial fibrillation. Europace. 2021 Oct 9;23(10):1528-1538. doi: 10.1093/europace/euab087. PMID 34279604
- [Result] Kim D, Yang PS, You SC, Sung JH, Jang E, Yu HT, Kim TH, Pak HN, Lee MH, Lip GYH, Joung B. Treatment timing and the effects of rhythm control strategy in patients with atrial fibrillation: nationwide cohort study. BMJ. 2021 May 11;373:n991. doi: 10.1136/bmj.n991. PMID 33975876
- [Result] Thomas L, Abhayaratna WP. Left Atrial Reverse Remodeling: Mechanisms, Evaluation, and Clinical Significance. JACC Cardiovasc Imaging. 2017 Jan;10(1):65-77. doi: 10.1016/j.jcmg.2016.11.003. PMID 28057220
- [Result] Wylie JV Jr, Peters DC, Essebag V, Manning WJ, Josephson ME, Hauser TH. Left atrial function and scar after catheter ablation of atrial fibrillation. Heart Rhythm. 2008 May;5(5):656-62. doi: 10.1016/j.hrthm.2008.02.008. Epub 2008 Feb 8. PMID 18452866
- [Result] Soulat-Dufour L, Lang S, Addetia K, Ederhy S, Adavane-Scheuble S, Chauvet-Droit M, Jean ML, Nhan P, Ben Said R, Kamami I, Issaurat P, Capderou E, Arnaud C, Boccara F, Lang RM, Cohen A. Restoring Sinus Rhythm Reverses Cardiac Remodeling and Reduces Valvular Regurgitation in Patients With Atrial Fibrillation. J Am Coll Cardiol. 2022 Mar 15;79(10):951-961. doi: 10.1016/j.jacc.2021.12.029. PMID 35272799
- [Result] January CT, Wann LS, Calkins H, Chen LY, Cigarroa JE, Cleveland JC Jr, Ellinor PT, Ezekowitz MD, Field ME, Furie KL, Heidenreich PA, Murray KT, Shea JB, Tracy CM, Yancy CW. 2019 AHA/ACC/HRS Focused Update of the 2014 AHA/ACC/HRS Guideline for the Management of Patients With Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2019 Jul 9;74(1):104-132. doi: 10.1016/j.jacc.2019.01.011. Epub 2019 Jan 28. No abstract available. PMID 30703431
- [Result] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Result] Asad ZUA, Yousif A, Khan MS, Al-Khatib SM, Stavrakis S. Catheter Ablation Versus Medical Therapy for Atrial Fibrillation: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Circ Arrhythm Electrophysiol. 2019 Sep;12(9):e007414. doi: 10.1161/CIRCEP.119.007414. Epub 2019 Aug 21. PMID 31431051
- [Result] Turagam MK, Musikantow D, Whang W, Koruth JS, Miller MA, Langan MN, Sofi A, Choudry S, Dukkipati SR, Reddy VY. Assessment of Catheter Ablation or Antiarrhythmic Drugs for First-line Therapy of Atrial Fibrillation: A Meta-analysis of Randomized Clinical Trials. JAMA Cardiol. 2021 Jun 1;6(6):697-705. doi: 10.1001/jamacardio.2021.0852. PMID 33909022
- [Result] Metzner A, Suling A, Brandes A, Breithardt G, Camm AJ, Crijns HJGM, Eckardt L, Elvan A, Goette A, Haegeli LM, Heidbuchel H, Kautzner J, Kuck KH, Mont L, Ng GA, Szumowski L, Themistoclakis S, van Gelder IC, Vardas P, Wegscheider K, Willems S, Kirchhof P. Anticoagulation, therapy of concomitant conditions, and early rhythm control therapy: a detailed analysis of treatment patterns in the EAST - AFNET 4 trial. Europace. 2022 Apr 5;24(4):552-564. doi: 10.1093/europace/euab200. PMID 34473249
- [Result] Lavee J, Onik G, Mikus P, Rubinsky B. A novel nonthermal energy source for surgical epicardial atrial ablation: irreversible electroporation. Heart Surg Forum. 2007;10(2):E162-7. doi: 10.1532/HSF98.20061202. PMID 17597044
- [Result] Cochet H, Nakatani Y, Sridi-Cheniti S, Cheniti G, Ramirez FD, Nakashima T, Eggert C, Schneider C, Viswanathan R, Derval N, Duchateau J, Pambrun T, Chauvel R, Reddy VY, Montaudon M, Laurent F, Sacher F, Hocini M, Haissaguerre M, Jais P. Pulsed field ablation selectively spares the oesophagus during pulmonary vein isolation for atrial fibrillation. Europace. 2021 Sep 8;23(9):1391-1399. doi: 10.1093/europace/euab090. PMID 33961027
- [Result] Reddy VY, Gerstenfeld EP, Natale A, Whang W, Cuoco FA, Patel C, Mountantonakis SE, Gibson DN, Harding JD, Ellis CR, Ellenbogen KA, DeLurgio DB, Osorio J, Achyutha AB, Schneider CW, Mugglin AS, Albrecht EM, Stein KM, Lehmann JW, Mansour M; ADVENT Investigators. Pulsed Field or Conventional Thermal Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2023 Nov 2;389(18):1660-1671. doi: 10.1056/NEJMoa2307291. Epub 2023 Aug 27. PMID 37634148
- [Result] Tops LF, Delgado V, Bertini M, Marsan NA, Den Uijl DW, Trines SA, Zeppenfeld K, Holman E, Schalij MJ, Bax JJ. Left atrial strain predicts reverse remodeling after catheter ablation for atrial fibrillation. J Am Coll Cardiol. 2011 Jan 18;57(3):324-31. doi: 10.1016/j.jacc.2010.05.063. PMID 21232671
- [Result] Schipper JH, Steven D, Luker J, Wormann J, van den Bruck JH, Filipovic K, Dittrich S, Scheurlen C, Erlhofer S, Pavel F, Sultan A. Comparison of pulsed field ablation and cryoballoon ablation for pulmonary vein isolation. J Cardiovasc Electrophysiol. 2023 Oct;34(10):2019-2026. doi: 10.1111/jce.16056. Epub 2023 Sep 8. PMID 37682001
- [Result] Urbanek L, Bordignon S, Schaack D, Chen S, Tohoku S, Efe TH, Ebrahimi R, Pansera F, Hirokami J, Plank K, Koch A, Schulte-Hahn B, Schmidt B, Chun KJ. Pulsed Field Versus Cryoballoon Pulmonary Vein Isolation for Atrial Fibrillation: Efficacy, Safety, and Long-Term Follow-Up in a 400-Patient Cohort. Circ Arrhythm Electrophysiol. 2023 Jul;16(7):389-398. doi: 10.1161/CIRCEP.123.011920. Epub 2023 May 31. PMID 37254781